CLINICAL TRIAL: NCT03050359
Title: A Randomized Double-Blind, Double-Dummy, Phase 3 Study to Evaluate the Efficacy and Safety of Oral TAK-438 20 mg Compared to Lansoprazole 30 mg Once- or Twice-Daily in the Treatment of Endoscopically Confirmed Duodenal Ulcer Subjects With or Without Helicobacter Pylori Infection
Brief Title: Comparison of TAK-438 (Vonoprazan) to Lansoprazole in the Treatment of Duodenal Ulcer Participants With or Without Helicobacter Pylori Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-438_304; U1111-1139-0293 (Registry Identifier: WHO); CTR20170104 (Registry Identifier: CFDA)
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Results first posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-05

CONDITIONS: Duodenal Ulcer
Keywords: Drug therapy; Gastrointestinal Diseases; Digestive System Diseases; Lansoprazole; Anti-Ulcer Agents; Gastrointestinal Agents; Proton Pump Inhibitors; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Duodenal Ulcer; Gastrointestinal Diseases; Digestive System Diseases | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAK-438 20 mg (Experimental): H. pylori negative (HP -) participants: TAK-438 20 mg, tablets, orally, once daily (QD) and lansoprazole placebo-matching capsules, orally, QD for up to 6 weeks. H. pylori positive (HP +) participants: TAK-438 20 mg, tablets, orally, twice daily (BID) and lansoprazole placebo-matching capsules, orally, BID for first 2 weeks along with Bismuth-Containing Quadruple Therapy followed byTAK-438 20 mg, tablets, orally, QD and lansoprazole placebo-matching capsules, orally, QD for up to 4 weeks.
  Interventions: Drug: TAK-438; Drug: Lansoprazole Placebo; Drug: Bismuth-Containing Quadruple Therapy
- Lansoprazole 30 mg (Experimental): H. pylori negative (HP -) participants: lansoprazole 30 mg, capsules, orally, QD and TAK-438 placebo-matching tablets, orally, QD for up to 6 weeks. HP + participants: lansoprazole 30 mg, capsules, orally, BID and TAK-438 placebo-matching tablets, orally, BID for first 2 weeks along with Bismuth-Containing Quadruple Therapy followed by lansoprazole 30 mg, capsules, orally, QD and TAK-438 placebo-matching tablets, orally, BID for up to 4 weeks.
  Interventions: Drug: Lansoprazole; Drug: TAK-438 Placebo; Drug: Bismuth-Containing Quadruple Therapy

INTERVENTIONS:
Drug: TAK-438 — TAK-438 tablets
  Other Names: Vonoprazan
  Arms: TAK-438 20 mg
Drug: Lansoprazole — Lansoprazole capsules
  Other Names: Prevacid
  Arms: Lansoprazole 30 mg
Drug: TAK-438 Placebo — TAK-438 placebo-matching tablets.
  Arms: Lansoprazole 30 mg
Drug: Lansoprazole Placebo — Lansoprazole placebo-matching capsules
  Arms: TAK-438 20 mg
Drug: Bismuth-Containing Quadruple Therapy — 1 g Amoxicillin, 500 mg clarithromycin and 600 mg bismuth potassium citrate/bismuth tripotassium dicitrate, twice daily (BID).

SUMMARY:
The purpose of this study is to demonstrate the non-inferior efficacy of TAK-438 versus lansoprazole in the treatment of participants with duodenal ulcer.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-438. TAK-438 is being tested to treat people who have duodenal ulcers and also may or may not have Helicobacter pylori (HP) infection. This study will look at duodenal ulcer healing and also the elimination of HP in people who take TAK-438 versus lansoprazole. The study will enroll approximately 530 patients.

Participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which remained undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* TAK-438 20 mg
* Lansoprazole 30 mg

HP+ participants will be asked to take a TAK- 438 tablet and a lansoprazole capsule twice daily in conjunction with bismuth-containing quadruple therapy for 2 weeks, followed up by a TAK-438 tablet and a lansoprazole capsule once daily for up to 4 weeks. HP negative (HP-) participants will be asked to take a TAK-438 tablet and a lansoprazole capsule once daily for up to 6 weeks.

This multi-center trial will be conducted China, Korea and Taiwan. The overall time to participate in this study is up to 10 weeks. Participants will make multiple visits plus final visit at 2 weeks or 4 weeks after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has endoscopic evidence of active duodenal ulcer(s) (i.e., mucosal defects with white coating [including cases associated with blood coagulation as long as there is no active bleeding]) measuring 5 mm or larger in longest diameter within 14 days prior to randomization.

Exclusion Criteria:

1. Has received TAK-438 in a previous clinical study or as a therapeutic agent.
2. Has a history or clinical manifestations of significant central nervous system (CNS), cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urological, endocrine or hematological disease that, in the opinion of the investigator, would confound the study results or compromise participant safety.
3. Has been treated with Helicobacter pylori eradication therapy within 30 days prior to study treatment.
4. Has a diagnosis of duodenal malignancy or a duodenal ulcer whose morphology suggested malignancy as evident by endoscopy within 14 days prior to randomization.
5. Is suspected of having acute gastro-duodenal mucosal lesions (AGDML) as evident by endoscopy within 14 days prior to randomization.
6. Has a linear ulcer (including a linear ulcer scar) that has been confirmed as evident by endoscopy within 14 days prior to randomization.
7. Has active postoperative (eg, endoscopic mucosal resection / endoscopic submucosal dissection) ulcer(s) as confirmed by endoscopy within 14 days prior to randomization.
8. Has gastric ulcer that has been confirmed by endoscopy within 14 days prior to randomization.
9. Has ulcers for which medical therapy alone is not indicated (eg, perforation, pyloric stenosis, duodenal stenosis, major bleeding).
10. Has undergone therapeutic upper gastrointestinal (GI) endoscopic therapy (eg, endoscopic hemostasis or excision including biopsy) within 30 days prior to visit 1.
11. Has Zollinger-Ellison syndrome or gastric acid hypersecretion or those with a history of gastric acid hypersecretion.
12. Has undergone major surgical procedures within 30 days prior to Visit 1 or are scheduled to undergo surgical procedures that may affect gastric acid secretion (eg, abdominal surgery, vagotomy or craniotomy).
13. Has a history of malignancy or was treated for malignancy within 5 years before the start of the visit 1 (the participant may be included in the study if he/she has cured cutaneous basal cell carcinoma or cervical carcinoma in situ).
14. Has a known acquired immunodeficiency syndrome (AIDS) or hepatitis infection, including hepatitis virus carriers (hepatitis B surface-antigen [HBsAg] - or hepatitis C virus (HCV)-antibody-positive) (the participant may be included in the study if he/she is HCV-viral load-RNA-negative).
15. Laboratory tests performed prior to randomization revealed any of the following abnormalities in the participant:

    1. Creatinine levels: >2 mg/dL (>177 μmol/L).
    2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST), or total bilirubin levels: > upper limit of normal (ULN).
16. Has hypersensitivity to TAK-438, proton pump inhibitors (PPIs), bismuth, clarithromycin, or amoxicillin. Skin testing may be performed according to local standard practice (for HP+ participants only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (81):
- China (53):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Yijishan hospital of Wan nan Medical college, Wuhu, Anhui
  - Beijing Chao Yang Hospital, Beijing, Beijing Municipality
  - The General Hospital of People's Armed Police Forces China, Beijing, Beijing Municipality
  - The Central Hospital of China Aerospace Corporation, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tong Ren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing,P.R., Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fuzhou General Hospital of Nanjing Military Area Command of Chinese PLA, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhangzhou Hospital, Zhangzhou, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Haikou People's Hospital, Haikou, Hainan
  - Shiyan Taihe Hospital, Shiyan, Hebei
  - The 2nd Xiangya Hospital Central South University, Changsha, Hu'nan
  - Chenzhou No.1 People's Hospital, Chenzhou, Hu'nan
  - Changsha Central Hospital, Yuhua, Hu'nan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Union Hospital of Tongji Medical College of Huazhong Science and Techology University, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Wuhan General Hospital of Guangzhou Military, Wuhan, Hubei
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Wuxi 4th People's Hospital, Wuxi, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - Jiangxi Nanchang 3rd Hospital, Nanchang, Jiangxi
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Jilin 4th People'S hospital, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Jilin central Hospital, Jilin, Jilin
  - Jilin Siping Central Hospital, Siping, Jilin
  - General Hospital of Shenyang Military Region, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia Hui
  - People's Hospital of Qinghai Province, Xining, Qinghai
  - The 2nd Hospital of Xi An Jiaotong University, Xi'an, Shan'xi
  - Ruijin Hospital, Shanghai Jiaotong Uni. School of Med., Huangpu Qu, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Affiliated General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical College, Kunming, Yun'nan
  - 1st Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
- Philippines (6):
  - Cebu Doctors University Hospital, Cebu City
  - St. Luke's Medical Center Global City, City of Taguig
  - De La Salle University Medical Center, Dasmarinas City, Cavite
  - Davao Doctors Hospital, Davao City
  - West Visayas State University Medical Center, Iloilo City
  - Philippine General Hospital, Manila
- South Korea (17):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - The Catholic University of Korea, Bucheon St. Mary s Hospital, Bucheon-si, Gyeonggi-do
  - Hanyang Univerisy Guri Hospital, Guri-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Wonkwang University Hospital, Iksan-si, Jeollabuk-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
- Taiwan (5):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Hou X, Wang J, Du Q, Tian D, Hu N, Liu D, Zhou F, Xie L, Gu L, Kudou K, Zhang S. Efficacy and Safety of Vonoprazan-Based Quadruple Therapy for the Eradication of Helicobacter pylori in Patients with Peptic Ulcers: A Pooled Analysis of Two Randomized, Double-Blind, Double-Dummy, Phase 3 Trials. Biol Pharm Bull. 2024;47(8):1405-1414. doi: 10.1248/bpb.b24-00011. PMID 39085080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 52 investigative sites in China, Korea, and Taiwan from 05 April 2017 to 19 July 2019.
Pre-assignment Details: Participants with or without diagnosis of Helicobacter pylori (H. Pylori) Infection were enrolled and randomly assigned in 1:1 ratio to receive either TAK-438 20 mg or lansoprazole 30 mg along with matching placebo (to keep the blind).
Period: Overall Study
Arm/Group | TAK-438 20 mg | Lansoprazole 30 mg
Started | 265 | 268
Completed | 248 | 248
Not Completed | 17 | 20
Not completed — Randomized But Not Treated | 2 | 0
Not completed — Pretreatment Event/Adverse Event | 5 | 10
Not completed — Significant Protocol Deviation | 2 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Voluntary Withdrawal | 4 | 6
Not completed — Pregnancy | 1 | 0
Not completed — Reason Not Specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- TAK-438 20 mg: HP - participants: TAK-438 20 mg, tablets, orally, once daily (QD) and lansoprazole placebo-matching capsules, orally, QD for up to 6 weeks. HP + participants: TAK-438 20 mg, tablets, orally, twice daily (BID) and lansoprazole placebo-matching capsules, orally, BID for first 2 weeks along with Bismuth-Containing Quadruple Therapy followed byTAK-438 20 mg, tablets, orally, QD and lansoprazole placebo-matching capsules, orally, QD for up to 4 weeks.
- Lansoprazole 30 mg: HP - participants: lansoprazole 30 mg, capsules, orally, QD and TAK-438 placebo-matching tablets, orally, QD for up to 6 weeks. HP + participants: lansoprazole 30 mg, capsules, orally, BID and TAK-438 placebo-matching tablets, orally, BID for first 2 weeks along with Bismuth-Containing Quadruple Therapy followed by lansoprazole 30 mg, capsules, orally, QD and TAK-438 placebo-matching tablets, orally, BID for up to 4 weeks.
- Total: Total of all reporting groups
Arm/Group | TAK-438 20 mg | Lansoprazole 30 mg | Total
Number analyzed (Participants) | 265 | 268 | 533
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (12.18) | 41.4 (12.89) | 41.7 (12.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 92 | 191
  Male | 166 | 176 | 342
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 265 | 268 | 533
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 252 | 255 | 507
  Korea, Republic Of | 10 | 8 | 18
  Taiwan, Province Of China | 3 | 5 | 8
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 166.1 (8.21) | 167.1 (8.09) | 166.6 (8.16)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — Population: Number analyzed is the number of participants with data available for weight at Baseline.
  kilograms (kg)
    number analyzed (Participants) | 263 | 268 | 531
    (all) | 63.45 (12.342) | 64.00 (11.383) | 63.72 (11.860)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index=weight (kg)/[height (m)^2] Population: Number analyzed is the number of participants with data available for BMI at Baseline.
  kg/m^2
    number analyzed (Participants) | 263 | 268 | 531
    (all) | 22.87 (3.365) | 22.83 (3.181) | 22.85 (3.270)
Smoking Classification [Count of Participants; unit: Participants]
  The Participant Has Never Smoked | 164 | 165 | 329
  The Participant Is a Current Smoker | 86 | 84 | 170
  The Participant Is an Ex-smoker | 15 | 19 | 34
Consumption of Alcohol [Count of Participants; unit: Participants]
  Drink Everyday | 6 | 2 | 8
  Drink a Couple of Days Per Week | 20 | 21 | 41
  Drink a Couple of Days Per Month | 48 | 58 | 106
  Never Drink | 191 | 187 | 378
Consumption of Caffeine [Count of Participants; unit: Participants]
  Yes (More Than 5 Times Per Week) | 23 | 16 | 39
  No (Never Drink or Less Than 5 Times Per Week) | 242 | 252 | 494
History of H.pylori Eradication Therapy [Count of Participants; unit: Participants]
  Yes (Therapy Received Ever) | 16 | 5 | 21
  No (Never Receive Any Therapy) | 249 | 263 | 512
H. pylori Infection Status [Count of Participants; unit: Participants] — Participants were evaluated for the H.pylori infection by result of 13C Urea Breath Test. Participants with infection were categorized as positive. Participants without infection were categorized as negative. Population: Number analyzed is the number of participants with data available for H. pylori Infection status at Baseline.
  Participants
    number analyzed (Participants) | 263 | 267 | 530
    Positive | 226 | 229 | 455
    Negative | 37 | 38 | 75
Characteristics of Current Duodenal Ulcers (DU): Location [Count of Participants; unit: Participants] — Participants were categorized based on their location of ulcer. Population: Number analyzed is the number of participants with data available for location of ulcer at Baseline.
  Participants
    number analyzed (Participants) | 265 | 267 | 532
    Superior Part (Including Bulb) | 262 | 266 | 528
    Descending Part | 3 | 1 | 4
Characteristics of Current DU: Mean Number of Ulcers Found [Mean (Standard Deviation); unit: number of ulcers] — Population: Number analyzed is the number of participants with data available for number of ulcers found at Baseline.
  number of ulcers
    number analyzed (Participants) | 263 | 268 | 531
    (all) | 1.2 (0.48) | 1.3 (0.54) | 1.2 (0.51)
Characteristics of Current DU: Ulcer Morphology [Count of Participants; unit: Participants] — Participants were categorized based on the morphology (shape) of ulcer: circular, ellipsoidal or other.
  Participants
    Circular | 110 | 117 | 227
    Ellipsoidal | 109 | 107 | 216
    Other | 46 | 44 | 90
Characteristics of Current DU: Ulcer Size [Count of Participants; unit: Participants] — Participants were categorized based on the size of ulcer: minuscule (<5 mm), minor (>=5 mm/<10 mm), intermediate (>=10 mm/<=20 mm), large (>20 mm/<30 mm), giant (>=30 mm).
  Participants
    Minuscule (<5 mm) | 0 | 1 | 1
    Minor (>=5 mm/<10 mm) | 183 | 188 | 371
    Intermediate (>=10 mm/<=20 mm) | 81 | 78 | 159
    Large (>20 mm/<30 mm) | 1 | 0 | 1
    Giant (>=30 mm) | 0 | 1 | 1
History of DU: Time Since Onset of Current Ulcers [Median (Full Range); unit: days] — Time since onset of current ulcers is defined as time in days from enrolment up to the onset of current ulcer.
  days | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
Use of NSAIDs or Low-dose Aspirin at the Time of Ulcer Onset [Count of Participants; unit: Participants] — Participants who used the nonsteroidal anti-inflammatory drug (NSAID) were categorized as 'YES'. Participants who did not use the NSAID were categorized as 'NO'.
  Participants
    Yes | 1 | 2 | 3
    No | 264 | 266 | 530
History of DU: Type of Ulcers [Count of Participants; unit: Participants] — Participants were categorized based on the the type of ulcers: primary or recurrent
  Participants
    Primary | 230 | 227 | 457
    Recurrent | 35 | 41 | 76
Time Since Onset of Recurrent Ulcers [Mean (Standard Deviation); unit: days] — Time since onset of recurrent ulcers is defined as time in days from enrolment up to the onset of previous ulcer.
  days | 1149.3 (910.72) | 999.7 (828.57) | 1068.7 (859.12)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Endoscopically Confirmed Healing of Duodenal Ulcers
Description: Endoscopic healing was defined as the disappearance of all white coats associated with duodenal ulcers as confirmed endoscopically.
Time Frame: Week 4 or Week 6
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of the study drug. Overall number of participants analyzed were participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-438 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 254 | 255
percentage of participants | 96.9 [93.889 to 98.631] | 96.5 [93.406 to 98.374]
Statistical Analysis 1: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Test type: Non-Inferiority — If the lower bound of the 95% CI was ≥-6%, the DU healing rate for TAK-438 was considered to be noninferior to that seen with lansoprazole; Exact (Clopper-Pearson) = 0.4, 95% CI 2-sided [-2.998 to 3.791]

2. Secondary Outcome: Percentage of Helicobacter Pylori Infected (HP+) Participants With Successful HP Eradication After 4 or 6 Weeks of Treatment
Description: HP infection status was determined by ^13C Urea Breath Test (^13C-UBT). The urea breath test is used to detect infection with HP, a bacteria associated with stomach ulcers, by testing individual breath samples in a central laboratory.
Time Frame: 4 weeks post treatment (Up to 10 weeks)
Population: Participants from FAS, included all participants who were randomized and received at least 1 dose of the study drug with H pylori positive status at Baseline with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- TAK-438 20 mg: HP + participants: TAK-438 20 mg, tablets, orally, twice daily (BID) and lansoprazole placebo-matching capsules, orally, BID for first 2 weeks along with Bismuth-Containing Quadruple Therapy followed byTAK-438 20 mg, tablets, orally, QD and lansoprazole placebo-matching capsules, orally, QD for up to 4 weeks.
- Lansoprazole 30 mg: HP + participants: lansoprazole 30 mg, capsules, orally, BID and TAK-438 placebo-matching tablets, orally, BID for first 2 weeks along with Bismuth-Containing Quadruple Therapy followed by lansoprazole 30 mg, capsules, orally, QD and TAK-438 placebo-matching tablets, orally, BID for up to 4 weeks.
Arm/Group | TAK-438 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 211 | 204
percentage of participants | 91.5 [86.853 to 94.866] | 86.8 [81.330 to 91.093]
Statistical Analysis 1: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Test type: Non-Inferiority — If the lower bound of the 95% CI was ≥-10%, the HP eradication rate for TAK-438 was considered to be noninferior to that seen with lansoprazole; Exact (Clopper-Pearson) = 4.7, 95% CI 2-sided [-1.281 to 10.690]

3. Secondary Outcome: Percentage of Participants With Endoscopically Confirmed Healing of Duodenal Ulcer at Week 4
Description: Endoscopic healing is defined as the disappearance of all white coats associated with duodenal ulcers as confirmed endoscopically.
Time Frame: Week 4
Population: FAS included all participants who were randomized and received at least 1 dose of the study drug. Overall number of participants analyzed were participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-438 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 249 | 251
percentage of participants | 89.2 [84.617 to 92.731] | 88.4 [83.830 to 92.124]
Statistical Analysis 1: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Exact (Clopper-Pearson) = 0.7, 95% CI 2-sided [-4.901 to 6.319]

4. Secondary Outcome: Percentage of Participants With Posttreatment Resolution of Gastrointestinal Symptoms Associated With Duodenal Ulcer at Weeks 2 Through 6
Description: The percentage of participants with resolution of various gastrointestinal symptoms are reported as categories. Gastrointestinal symptoms included epigastric pain (postprandial, fasting, nocturnal), abdominal bloating, nausea/vomiting, heartburn and lack of appetite. The severity of subjective symptoms of erosive esophagitis were recorded as: none = 0, mild = 1, moderate = 2 or severe = 3.
Time Frame: Week 2 up to Week 6
Population: FAS included all participants who were randomized and received at least 1 dose of the study drug. Number analyzed is number of participants analyzed for the particular category (symptom).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-438 20 mg | Lansoprazole 30 mg
Number analyzed (Participants) | 263 | 268
percentage of participants
  Epigastric Pain (Postprandial): number analyzed (Participants) | 57 | 49
  Epigastric Pain (Postprandial) | 87.7 [76.321 to 94.917] | 91.8 [80.399 to 97.731]
  Epigastric Pain (Fasting/Nocturnal): number analyzed (Participants) | 132 | 141
  Epigastric Pain (Fasting/Nocturnal) | 91.7 [85.579 to 95.767] | 90.1 [83.902 to 94.465]
  Abdominal Bloating: number analyzed (Participants) | 48 | 63
  Abdominal Bloating | 83.3 [69.778 to 92.519] | 87.3 [76.503 to 94.355]
  Nausea/Vomiting: number analyzed (Participants) | 27 | 18
  Nausea/Vomiting | 85.2 [66.269 to 95.811] | 94.4 [72.706 to 99.859]
  Heartburn: number analyzed (Participants) | 28 | 22
  Heartburn | 100.0 [87.656 to 100.000] | 95.5 [77.156 to 99.885]
  Lack of Appetite: number analyzed (Participants) | 22 | 18
  Lack of Appetite | 90.9 [70.839 to 98.879] | 100.0 [81.470 to 100.000]
Statistical Analysis 1: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Epigastric Pain (Postprandial); Test type: Other; Difference in percentages = -4.1, 95% CI 2-sided [-15.579 to 7.344]
Statistical Analysis 2: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Epigastric Pain (Fasting/Nocturnal); Test type: Other; Difference in percentages = 1.6, 95% CI 2-sided [-5.230 to 8.422]
Statistical Analysis 3: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Abdominal Bloating; Test type: Other; Difference in percentages = -4.0, 95% CI 2-sided [-17.338 to 9.401]
Statistical Analysis 4: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Nausea/Vomiting; Test type: Other; Difference in percentages = -9.3, 95% CI 2-sided [-26.334 to 7.815]
Statistical Analysis 5: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Heartburn; Test type: Other; Difference in percentages = 4.5, 95% CI 2-sided [-4.159 to 13.250]
Statistical Analysis 6: Comparison: TAK-438 20 mg vs Lansoprazole 30 mg; Lack of Appetite; Test type: Other; Difference in percentages = -9.1, 95% CI 2-sided [-21.104 to 2.922]

ADVERSE EVENTS:
Time Frame: Up to Week 10 (Up to 6 weeks of treatment)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-438 20 mg | Lansoprazole 30 mg
All-Cause Mortality (participants affected / at risk) | 0/263 | 0/268
Serious Adverse Events (participants affected / at risk) | 1/263 | 3/268
Other Adverse Events (participants affected / at risk) | 162/263 | 113/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-438 20 mg (N=263) | Lansoprazole 30 mg (N=268)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-438 20 mg (N=263) | Lansoprazole 30 mg (N=268)
Upper respiratory tract infection (Infections and infestations) | 21 | 37
Pepsinogen test positive (Investigations) | 124 | 28
Pepsinogen I increased (Investigations) | 92 | 37
Blood gastrin increased (Investigations) | 97 | 20
Protein urine present (Investigations) | 20 | 11
Alanine aminotransferase increased (Investigations) | 12 | 17
Dysgeusia (Nervous system disorders) | 21 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT03050359/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT03050359/SAP_001.pdf